CLINICAL TRIAL: NCT05090059
Title: Myofascial Points Treatment With Focused Extracorporeal Shock Waves (f-ESW) for Plantar Fasciitis: an Open Label Randomized Clinical Trial
Brief Title: Myofascial Points Treatment With Focused Extracorporeal Shock Waves (ESW)
Acronym: ESW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 61902
Record Dates: First submitted 2021-09-06; First posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-09

CONDITIONS: Plantar Fasciitis; Myofascial Trigger Point Pain; Foot Injury
MeSH Terms: conditions — Fasciitis, Plantar; Myofascial Pain Syndromes; Foot Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lower limb myofascial trigger points f-ESWT group (Experimental): 3 total sessions, one per week, of focused extracorporeal shockwave treatment with a frequency of 5 Hz, an energy flux density of 0.05-0.167 mJ (millijoule)/mm2 administered on 3 or 4 myofascial points (identified based on Fascial Manipulation principles), 1500 shocks per point.
  Interventions: Device: Lower limb myofascial trigger points f-ESWT
- Plantar fascia insertion f-ESWT group (Active Comparator): 3 total sessions, one per week, of focused extracorporeal shockwave treatment, with a frequency of 5 Hz, an energy flux density of 0.32 mJ(millijoule)/mm2, for a total of 2000 shocks administered on the area of the painful heel on the medial calcaneal tubercle.
  Interventions: Device: Lower limb myofascial trigger points f-ESWT

INTERVENTIONS:
Device: Lower limb myofascial trigger points f-ESWT — 3 weekly sessions of focused Extracorporeal Shockwave treatment with a frequency of 5 Hz, an energy flux density of 0.05-0.167 mJ(millijoule)/mm2, administered on 3-4 myofascial lower limb trigger points (identified according to the approach of Fascial Manipulation), 1500 shocks per point.

SUMMARY:
Plantar fasciitis (PF) is a common cause of heel pain. Among the several conservative treatment options, Extracorporeal Shock Wave Therapy (ESWT) is considered the standard treatment.

Recent studies suggest that PF may be sustained by a myofascial impairment proximal to the pain area with a biomechanical disequilibrium of the entire lower limb and pelvis. Therefore, by combining the concepts of Fascial Manipulation and ESWT, the purpose of this open label randomized controlled clinical trial is to evaluate the effectiveness of the ESWT on myofascial trigger points of lower limb in a sample of subjects with PF.

Patients with PF were randomly assigned to an Experimental treatment Group (EG), treated with focused ESWT on myofascial points, and a Control Group (CG), treated with the focused ESWT traditional approach on the medial calcaneal tubercle.

Outcome measures included the Foot and Ankle Outcome Score (FAOS) and the Italian Foot Functional Index (17-iFFI).

The assessment was made before the first session(baseline-T1), immediately before the second session (T2), immediately before the third session (T3), at 1month (T4) and 4 months' follow-up (T5).

Thirty patients who satisfied inclusion and exclusion criteria were enrolled.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age,
* the presence of heel pain ≥ 3 months duration unresponsive to first-choice conservative treatments (non-steroidal anti-inflammatory and/or other analgesic drugs, exercise program, insoles),
* specialist diagnosis of plantar fasciitis confirmed with clinical examination,
* pain intensity ≥ 5 at the Visual Analog Scale (VAS)

Exclusion Criteria:

* previous ankle/foot fracture or surgery,
* previous ankle/foot infections,
* neurological deficits of the lower limbs,
* diagnosis or suspect of fibromyalgia,
* local steroid injection within the previous 3 months,
* diabetes mellitus,
* vascular diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Change in 17-Italian Foot Function Index (17-iFFI) | T1 (baseline - immediately before the first session); T2 (1 week - immediately before the second session); T3 (2 weeks - immediately before the third session); T4 (1 month follow-up); T5 (4 months follow-up)
  Self-administered questionnaire. It consists in 17 items divided into 3 subscales: pain (5 items), disability (9 items), and limitation of activity (3 items). The items are rated on a Visual Analogue Scale (VAS), from 0 to 10.
  A score is calculated for every subgroup of items, and then the final score is calculated by adding the subscale's scores and dividing the result by 170. The final percentage score is between 0% (best outcome) and 100% (worst outcome).
Change in Foot and Ankle Outcome Scale (FAOS) | T1 (baseline - immediately before the first session); T2 (1 week - immediately before the second session); T3 (2 weeks - immediately before the third session); T4 (1 month follow-up); T5 (4 months follow-up)
  Self-administered questionnaire. It consists of 42 items divided in 5 subscales: pain (9 items), other symptoms (7 items), function in activities of daily living (17 items), function in sports and recreation (5 items), and foot-and-ankle related quality of life (4 items).
  The questions are made to be answered with qualitative terms (None, Mild, Moderate, Severe, Extreme) or temporal terms (Never, Rarely, Sometimes, Often, Always) corresponding to a numeric value, from 0 to 4. The score for each subdomain as well as the total FAOS is then calculated and normalized to a 0-100 scale, where 0% is the worst outcome and 100% the best outcome. Then, a final, global percentage score, from 0% (worst outcome) to 100% (best outcome), is given.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurosciences, Physical and Rehabilitation Unit, University of Padova, Padua, Italy

IPD SHARING:
Plan to Share IPD: Undecided